CLINICAL TRIAL: NCT04546997
Title: Retinal Vascular Features in Ocular Blunt Trauma by Optical Coherence Tomography Angiography
Brief Title: Study of Retinal Vascular Changes After Ocular Blunt Trauma
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 1212/2019
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Ocular Injury
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ocular blunt trauma: Patients with previous ocular blunt trauma in one eye.
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography
- Control Group: Healthy fellow eyes without actual and previous ocular trauma
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography — Patients underwent non-invasive, fast, diagnostic imaging technique (optical coherence tomography angiography)

SUMMARY:
This study evaluates the retinal vascular features using optical coherence tomography angiography in patients that received ocular blunt trauma.

DETAILED DESCRIPTION:
To investigate, using optical coherence tomography angiography, early retinal vascular features 48 hours after ocular trauma and to detect their changes during 6 months' follow up.

The optical coherence tomography angiography represents a novel and noninvasive diagnostic technique that allows a detailed analysis of retinal vascular features.

ELIGIBILITY:
Inclusion Criteria:

* age older than 40 years
* diagnosis of previous ocular blunt trauma
* absence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* absence of significant lens opacities, low-quality OCT and OCT-A images.

Exclusion Criteria:

* age younger than 40 years
* absence of previous ocular blunt trauma
* presence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* presence of significant lens opacities, low-quality OCT and OCT-A images.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participans were older than 40 years with diagnosis of previous ocular blunt trauma. They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal vessel density in patients after ocular blunt trauma during 6 months's follow up | Six months
  To evaluate the changes in retinal vessel density in 18 patients, at baseline and 1, 3, 6 months after ocular blunt trauma, using optical coherence tomography angiography.
  The parameter analyzed by optical coherence tomography angiography was: retinal vessel density

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, MD, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy